CLINICAL TRIAL: NCT06777875
Title: COMT and OPRM1 Polymorphisms and Their Effect on Post-Operative Pain in Children Undergoing Orthopedic, Abdominal, Thoracic, and Plastic Surgeries.
Brief Title: COMT and OPRM1 Polymorphisms and Their Effect on Post-Operative Pain in Children
Status: Recruiting | Type: Observational
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Roland Kaddoum, Principal Investigator, American University of Beirut Medical Center
Other Study IDs: BIO-2024-0365
Record Dates: First submitted 2025-01-09; First posted 2025-01-16 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Pain; Genetic Change; Children, Only
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous whole blood (2 mL) will be sampled into coded Ethylenediaminetetraacetic acid (EDTA) tubes at the time of study enrollment and stored at -80°C. Samples will be obtained during the insertion of the IV in preparation for anesthesia or as left over from blood withdrawn for complete blood count (CBC) in an EDTA purple tube. Genomic DNA will be purified from each blood using a Qiagen kit according to the manufacturer's instructions. Four Catechol-O-methyltransferase (COMT) single-nucleotide polymorphisms (SNPs) (rs6269, rs4633, rs4818, rs4680 and the rs179971 variant.).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to investigate whether the A118G single-nucleotide polymorphism (SNP) in the mu-opioid receptor1(OPRM1) and Catechol-O-methyltransferase (COMT) SNPs influence postoperative pain scores in children between the ages of 8 and 18 undergoing orthopedic, abdominal, thoracic, and plastic surgeries.

The main question[s] it aims to answer [is]:

Do OPRM1 and COMT SNPs influence postoperative pain scores in children between the ages of 8 and 18 undergoing orthopedic, abdominal, thoracic, and plastic surgeries?

Participants will be assessed for their pain scores, sedation level, the amount of postoperative analgesics received, duration of their stay in the post-anesthesia care unit, and toxicity.

DETAILED DESCRIPTION:
Inadequately treated pain in children undergoing surgery is a major concern for health providers. Recent evidence indicates that pain sensitivity differs among races and ethnicities and genetic makeup. Catechol-O-methyltransferase (COMT) polymorphisms (rs6269, rs4633, rs4818 and rs4680) which are inherited together in different phenotypes influence clinical presentations and responses to pain.

A118G single-nucleotide polymorphism (SNP) in the mu-opioid receptor1 (OPRM1) gene is associated with differences in pain perception and opioid requirements. The effect of genome variations in the COMT gene and in the OPRM1 on postoperative pain perception and morphine analgesia in children needs further exploration. The main objective of this study was to investigate whether the OPRM1 and COMT SNPs influence postoperative pain scores in children between the ages of 8 and 18 undergoing orthopedic, abdominal, thoracic, and plastic surgeries. Secondary objective includes assessing whether OPRM1 and COMT SNPs influence postoperative sedation score, intraoperative and postoperative opioid requirements, length of stay in the post anesthesia care unit (PACU), and signs of respiratory depression (RD) and postoperative nausea and vomiting (PONV).

Methodology: A prospective cohort genotype-blinded observational study will be conducted. A convenience sample of 200 children between the ages of 8-18 undergoing orthopedic, abdominal, thoracic, and plastic surgeries will be recruited from the American University of Beirut Medical Center (AUBMC). The primary outcome of the study is the post operative pain score in PACU.

Secondary outcomes include the postoperative sedation score, intraoperative and postoperative opioid requirements, length of stay in the PACU, and signs of RD and PONV. To test the hypothesis that COMT and OPRM1 SNPs are associated with postoperative analgesia outcomes in children, SPSS version 29 will be used. Allelic and genotype frequencies will be examined by the Hardy-Weinberg equilibrium (HWE) test. To analyze the association between the different genetic variations and the outcomes, bivariate analysis will be performed. Variables measured over time will be compared between the groups using an exploratory mixed model analysis. Time to first post-operative opioid requirement will be analyzed using the survival analysis Kaplan Meier curve. Such understanding will pave the way for individual tailoring and optimization of pain assessment and management in children undergoing orthopedic, abdominal, thoracic, and plastic surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* All children 8 years to 18 years
* Undergoing orthopedic, abdominal, thoracic, and plastic surgeries
* American Society of Anesthesiologists classification (ASA) I-II-III

Exclusion Criteria:

* Children with schizoid personality disorders, phobias, and anxiety
* Patients with neuropathic pain associated with surgeries requiring surgical treatment.
* Children presented with all types of depressive disorders, atypical bipolar disorder, or a suspicion of substance abuse.
* American Society of Anesthesiologists classification (ASA) ≥IV
* All patients receiving regional anesthesia, local blocks, epidural and caudal blocks.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children between the ages of 8-18 undergoing orthopedic, abdominal, thoracic, and plastic surgeries will be recruited from the American University of Beirut Medical Center (AUBMC).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-01-13 (Estimated); Study Completion 2027-01-13 (Estimated)

PRIMARY OUTCOMES:
Pain scores | Until discharge from PACU (about 3 hours)
  Pain scores measured using the Numerical Rating Scale (NRS) (ranging from 0 to 10, with 0 no pain and 10 worst pain)

SECONDARY OUTCOMES:
Postoperative sedation | Until discharge from PACU (about 3 hours)
  Postoperative sedation measured using the Richmond Agitation Sedation Scale (RASS) (ranging from -5 to +4, with -5 unarousable and +4 combative)
Use of intraoperative and post-operative opioids | Until discharge from PACU (about 3 hours)
  Use of intraoperative and post-operative opioids (Yes/No)
Length of post-anesthesia care unit (PACU) stay | Until discharge from PACU (about 3 hours)
  Length of post-anesthesia care unit (PACU) stay measured in hours
Postoperative respiratory depression | Until discharge from PACU (about 3 hours)
  Postoperative respiratory depression (Yes/No)
Postoperative nausea and vomiting | Until discharge from PACU (about 3 hours)
  Postoperative nausea and vomiting (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Roland Kaddoum, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- Roland Kaddoum, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No